CLINICAL TRIAL: NCT00230789
Title: A Multicenter, Multiphase, Single Arm, Open Label Study To Evaluate The Effects Of Tolterodine ER In Conjunction With Behavioral Intervention On Subject Satisfaction And Over- Active Bladder Symptoms (Urgency Urinary Incontinence (UUI), Urgency, Frequency) In Overactive Bladder Subjects Who Were Dissatisfied With Their Most Recent Antimuscarinic OAB Medication Therapy.
Brief Title: Effect Of Detrol LA With Behavioral Intervention In Overactive Bladder Subjects Dissatisfied With Recent OAB Medication.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6121146
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Tolterodine Tartrate

INTERVENTIONS:
Drug: Tolterodine ER 4 mg QD
Behavioral: OAB Patient Behavioral Training Material

SUMMARY:
To evaluate the effect of tolterodine ER in conjunction with behavioral intervention on subject satisfaction in OAB subjects who were dissatisfied with their most recent antimuscarinic OAB medication therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects greater than or equal to 18 years of age
* Overactive bladder symptoms for at least 3 months
* Previously treated with antimuscarinic OAB medications

Exclusion Criteria:

* Participation in any professionally coached sessions (RN, NP, PA or PT) teaching behavioral interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417
Dates: Start 2005-10; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Subject satisfaction with treatment at week 16: Percentage of subjects reporting satisfaction with their current OAB treatment using the Patient Perception of Treatment Satisfaction Question

SECONDARY OUTCOMES:
Percentage of subjects reporting satisfaction (including 'very satisfied' and 'a little satisfied') with their current OAB treatment measured by Patient Perception of Treatment Satisfaction
Percent subjects changed dissatisfied(including'very dissatisfied'and'a little dissatisfied')with OAB week 8 to satisfied(including'very satisfied' and'a little satisfied')with OAB week 16 measured by Patient Perception of Treatment Satisfaction Question
Change in mean number of urgency urinary incontinence episodes at weeks 4, 8, 12 and 16 compared with baseline
Change in mean number of urgency episodes per day at weeks 4, 8, 12 and 16 compared with baseline (Urgency episode defined as micturition episodes associated with Urinary Sensation Scale rating of greater than or equal to 3).
Change in daily urgency micturition rating at weeks 4,8,12 and 16 compared with baseline:Change in mean and sum of Urinary Sensation Scale rating per day
Change in mean number of micturition episodes per 24 hour period and per nocturnal period at weeks 4, 8, 12 and 16 compared with baseline. Means will be based on five dairy days. The following micturition episode parameters will be assessed:
Total micturitions: total number of micturition episodes per time period (24 hour or nocturnal)
OAB micturition: Number of OAB mictruition episodes per time period (24 hour or nocturnal). OAB micturition defined as number of micturition episodes associated with Urinary Sensation Scale ratting of greater than or equal to 3
Severe OAB micturitions in subjects with severe OAB micturition at baseline: Number of severe OAB micturition episodes per time period (24 hour or nocturnal).
Severe OAB micturition episodes defined as number of micturitions associated with a Urinary Sensation Scale rating of greater than or equal to 4
Change in Patient Perception of Bladder Condition (PPBC) at weeks 8 and 16 compared with baseline
Change in Patient Perception of Urgency Scale (PPUS) at weeks 8 and 16 compared with baseline
Change in total Health Related Quality of Life (HRQoL) for Overactive Bladder Questionnaire (OAB-q) and change in scores for each individual domain (symptom bother, coping, concern, sleep, and social function) at weeks 8 and 16 compared with baseline
Reasons for treatment withdrawal.
Adverse events during the 16 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (51):
- United States (51):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Sun Lakes, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Buena Park, California
  - Pfizer Investigational Site, Mission Viejo, California
  - Pfizer Investigational Site, Modesto, California
  - Pfizer Investigational Site, Oceanside, California
  - Pfizer Investigational Site, Paramount, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Wheat Ridge, Colorado
  - Pfizer Investigational Site, Hallandale, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Wellington, Florida
  - Pfizer Investigational Site, Woodstock, Georgia
  - Pfizer Investigational Site, Libertyville, Illinois
  - Pfizer Investigational Site, Mattoon, Illinois
  - Pfizer Investigational Site, Newton, Kansas
  - Pfizer Investigational Site, Milford, Massachusetts
  - Pfizer Investigational Site, Manchester, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Westhampton, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Endwell, New York
  - Pfizer Investigational Site, Garden City, New York
  - Pfizer Investigational Site, Poughkeepsie, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Greensboro, North Carolina
  - Pfizer Investigational Site, Hickory, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Canton, Ohio
  - Pfizer Investigational Site, Zanesville, Ohio
  - Pfizer Investigational Site, Norman, Oklahoma
  - Pfizer Investigational Site, Abington, Pennsylvania
  - Pfizer Investigational Site, Bala-Cynwyd, Pennsylvania
  - Pfizer Investigational Site, Camp Hill, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Williamsport, Pennsylvania
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Simpsonville, South Carolina
  - Pfizer Investigational Site, Bartlett, Tennessee
  - Pfizer Investigational Site, Johnson City, Tennessee
  - Pfizer Investigational Site, New Tazewell, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Provo, Utah
  - Pfizer Investigational Site, Mountlake Terrace, Washington
  - Pfizer Investigational Site, Spokane, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6121146&StudyName=Effect+Of+Detrol+LA+with+Behavioral+Intervention+In+Overactive+Bladder+Subjects+Dissatisfied+with+Recent+OAB+Medication%2E